CLINICAL TRIAL: NCT06372743
Title: A Dual-centre, Two-arm, Open-label Randomized Controlled Trial Comparing an Integrated Collaborative Nurse-led Physician-supported Multimorbid Chronic Kidney Disease Care Model Versus Physician-led Care (INTEGREAT-CKD)
Brief Title: Nurse-led Physician-supported Care for Patients With Chronic Kidney Disease and Multimorbidity
Acronym: INTEGREATCKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandra Hospital (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alex Hospital
Record Dates: First submitted 2023-10-30; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This study is a dual-centre two-arm, open-label randomized controlled trial (RCT). Patients are randomized with a one-to-one allocation into two parallel groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control arm: Patients will be assigned to a consultation model of CKD care which consists of clinic reviews by a nephrologist, which is as per current standard of care. The frequency of reviews, which is at the discretion of the nephrologist, is typically scheduled at 4 to 6 monthly intervals. Each consultation lasts an average of 10 to 15 minutes.
- INTEGREAT-CKD Intervention (Experimental): Intervention arm: Patients will be assigned to a consultation model of CKD care which consists of 30-minute clinic reviews led by an advanced practice nurse (APN), with both on-site and remote support from a nephrologist, at 3 monthly intervals. Patients will be required to monitor certain clinical parameters (one of or a combination of blood pressure, glucose trend or weight trend) between clinic reviews, tapping on a telehealth platform for transmission of data to an assigned community-based nurse, who will provide oversight of these readings, with regular escalation to the APN/nephrologist. The on-site remote support, in the form of telehealth monitoring, will be concurrent between clinic consults, with frequency of monitoring individualized as per patient's needs.
  Interventions: Other: INTEGREAT-CKD Intervention

INTERVENTIONS:
Other: INTEGREAT-CKD Intervention — The participant is reviewed once in 12 weeks by a CKD-trained APN, during a 30-minute timeslot, an extended duration compared to the timeslot of 10 to 15 minutes that routinely is designated for a recurrent review of a CKD patient in any restructured hospital in Singapore. The review consists of a 15-minute medical review centred on a discussion of the biochemical reports and clinical data relevant to CKD management, and educating on CKD knowledge and lifestyle modification.
  Patients self-report the monitored parameters to a community-based nurse through a telehealth AI-based platform. The APN oversees monitoring the community-based parameters and titration of appropriate medications. The APNs have received a Master's in Nursing, with training that is primarily centred on generalist-led care, with additional clinical training in CKD management. They are supported with protocols to detect anomalies in blood pressure trends, glycemia ranges, and abnormalities in fluid status.
  Arms: INTEGREAT-CKD Intervention

SUMMARY:
Chronic kidney disease (CKD) is a prevalent chronic disease and is often intertwined with the management of cardiovascular disease and the optimization of metabolic risk factors. In light of steeply rising rates of end-stage kidney disease (ESKD) and increased healthcare resource utilization by CKD patients, the investigators propose that the role of nurses could be expanded to support the care of CKD patients in the community.

A total of 220 patients will be randomized (1:1) to the intervention or control groups (usual care). The intervention entails enrolment into a nurse-led, physician-supported programme (INTEGREAT-CKD), comprising outpatient consultations and community-based ambulatory monitoring and counselling primarily driven by CKD-trained advanced practice nurses (APNs) and healthcare professionals conducted over 6 months. Patient-reported outcomes like health-related quality of life (HRQOL), as measured by EQ-5D and KDQOL, CKD self-management score and CKD health literacy will be assessed at baseline and after 6 months. The primary outcome is CKD self-management. Other secondary outcomes to be assessed and tracked including achievement of clinical targets relevant to slowing down CKD progression, attainment of CKD best practice guidelines as specified in the KDIGO CKD Evaluation and Management guidelines 2020.

DETAILED DESCRIPTION:
Study objectives:

1. To evaluate if a nurse-led model of care (INTEGREAT-CKD), in comparison to the standard of care (physician-led care), improves self-management skills, quality of life, and health literacy in patients with advanced CKD.
2. To assess if a nurse-led physician-supported consultation model of care, in comparison to the standard of care, optimizes the attainment of clinical targets following CKD best practice guidelines.
3. To assess if health resource utilization is cost-effective for complex CKD patients cared for by a nurse-led physician-supported consultation model of care compared to the standard of care.

Study design This study is a dual-centre two-arm, open-label randomized controlled trial (RCT). Patients are randomized with a one-to-one allocation into two parallel groups. Participants with advanced CKD referred to the tertiary institutions are randomized to either the control group (physician-led standard of care consultation model) or the experimental (intervention) group, which consists of enrolment in the INTEGREAT-CKD programme. INTEGREAT-CKD is a six-month programme consisting of an outpatient nurse-led consultation model, delivered by a team of CKD-trained Advanced Practice Nurses (APNs) and community-based nurses. Participants are reviewed in person at a 3-monthly interval by a CKD-trained APN independently. The CKD-trained APN's practice is supported by adherence to a protocol-based and algorithmic set of guidelines co-written by the CKD-trained APN and nephrologist for the main clinical aspects of CKD care. Each clinic session is allocated an extended duration of 30 minutes to educate patients on CKD-related medical knowledge, targeted lifestyle modification, and self-management skills. Questionnaires to determine patient's health literacy, self-management skills, and quality of life are assessed at the beginning and end of the study.

Setting:

The study will be conducted across two tertiary hospitals, Alexandra Hospital (AH) and National University Hospital (NUH), located in the western cluster of Singapore. Both hospitals are tertiary healthcare institutions that receive outpatient nephrology consult referrals, including consultation about CKD management, from within the institutions and primary healthcare sector within the western cluster.

Population and Sample:

The investigators plan to implement the envisioned intervention right from when CKD patients are referred to a nephrologist in one of the two institutions. Care received from this point onwards can significantly shape the course of a CKD patient's care journey.

Study Intervention Patients allocated to the intervention group will receive the nurse-led care (INTEGREAT-CKD), which comprises of the following components. Every recruited participant will be reviewed in person by a CKD-trained APN in the clinic on a 3-monthly basis for optimization of the medical management of CKD. Every patient is designated a 30-minute timeslot, an extended duration compared to the timeslot of 10 to 15 minutes that routinely is designated for a recurrent review of a CKD patient in any restructured hospital in Singapore. The 30-minute timeslot starts with a 15-minute medical review centred on a discussion of the biochemical reports and clinical data relevant to CKD management. The subsequent 15-minute time slot will be dedicated to educating patients on improving their knowledge of CKD, including the importance of optimizing clinical parameters that influence CKD progression.

Patients will be placed on community-based and monthly monitoring of clinical parameters relevant to CKD progression. Patients will self-report the monitored parameters to a community-based nurse through a telehealth platform.

Clinical parameters that are out of range will be escalated to the CKD-trained APN, who oversees the monitoring of the community-based monitored parameters and titration of appropriate medications.

Control group Patients assigned to the control group receive the usual standard of care at most specialist outpatient clinics in any tertiary restructured hospital in Singapore. They are not routinely scheduled to receive nurse-led CKD care - management by a CKD-trained APN and community-based monitoring of clinical parameters

Recruitment procedure CKD patients in Alexandra Hospital and National University Hospital who fulfill the study's inclusion criteria will be recruited for participation in the study. They may be recruited from the inpatient wards or outpatient clinics by a member of the research team. After providing written consent, the participants will be randomized to the intervention or control groups.

ELIGIBILITY:
Inclusion Criteria :

* Adults aged 21 years and above AND diagnosed with
* CKD Stages 3B and above (defined as estimated GFR less than or equal to 44 mL/min/1.73m2 with evidence of kidney damage) AND diagnosed with
* one or more of the following sub-optimally managed parameters pertaining to blood pressure control OR, glycemic control OR fluid status management.

Exclusion criteria:

* Pregnancy
* End stage kidney disease
* Enrolment in any structured outpatient-based or community-based CKD program for at least six months prior to or during the period of enrolment in the study.
* Dementia and/or cognitive impairment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic Kidney Disease Self-Management (CKD-SM) Questionnaire | 24 weeks from participants' date of enrollment
  Patients will be scored based on their questionnaire responses and the primary outcome is the improvement in the CKD-SM score. Baseline scoring is done during enrolment.

SECONDARY OUTCOMES:
Secondary outcome | 24 weeks from participants' date of enrollment
  (a) An achievement of clinical targets relevant to slowing down CKD progression:
  a. Individualised blood pressure target achieved depending on clinical profile: i. CKD, non-diabetic with proteinuria: < 140/80mmHg ii. CKD, diabetic with proteinuria: < 130/80 b. Target glycemia control: HbA1c lower than 8% c. Achievement and maintenance of euvolemia (individualized target weight that reflects euvolemia) (b) CKD best practice guidelines as specified in the KDIGO CKD Evaluation and Management guidelines
  a. Achievement of target biochemical indices related to optimization of CKD care: i. Mineral bone disease (CKD-MBD)
  1. Serum phosphate and serum calcium within normal ranges
  2. Serum parathyroid hormone to be maintained at approximately 2-9 times the upper normal limit for the assay{, #282} ii. Anemia
  1. Serum haemoglobin 10.5-11.5 g/dL (c) An improvement in the 30-day readmission (d) A reduction in the incidence of emergency department visits

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Zhen Hong, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stanifer JW, Von Isenburg M, Chertow GM, Anand S. Chronic kidney disease care models in low- and middle-income countries: a systematic review. BMJ Glob Health. 2018 Apr 1;3(2):e000728. doi: 10.1136/bmjgh-2018-000728. eCollection 2018. PMID 29629191
- [Result] Davis KM, Eckert MC, Hutchinson A, Harmon J, Sharplin G, Shakib S, Caughey GE. Effectiveness of nurse-led services for people with chronic disease in achieving an outcome of continuity of care at the primary-secondary healthcare interface: A quantitative systematic review. Int J Nurs Stud. 2021 Sep;121:103986. doi: 10.1016/j.ijnurstu.2021.103986. Epub 2021 May 27. PMID 34242979